CLINICAL TRIAL: NCT07186439
Title: Pulmonary Hypertension Screening in Scleroderma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Sayed Abdalazeaz, Resident at department chest diseas and tuberculosis, Assiut University
Other Study IDs: PHTN in scleroderma
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PHTN in Scleroderma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Screening for pulmonary hypertension in scleroderma patients

DETAILED DESCRIPTION:
Scleroderma is a heterogenous connective tissue disorder characterized by fibrosis of the skin, with or without internal organ involvement. The aetiology of scleroderma may involve both environmental and genetic factors. Abnormalities involving the immune system, vascular tissue and extracellular matrix have been demonstrated.

One of the major cause of mortality in patients with scleroderma is pulmonary arterial hypertension (PAH). International recommendations advise annual screening for the early detection of PAH in asymptomatic patients with scleroderma.

scleroderma is group 1 in clinical classification of pulmonary hypertension Pulmonary hypertension (PH) is a haemodynamic condition characterised by elevation of mean pulmonary arterial pressure (mPAP) >20 mmHg, assessed by right heart catheterisation. Pulmonary arterial wedge pressure (PAWP) and pulmonary vascular resistance (PVR) distinguish pre-capillary PH (PAWP ≤15 mmHg, PVR >2 Wood Units (WU)), isolated post-capillary PH (PAWP >15 mmHg, PVR ≤2 WU) and combined post- and pre-capillary PH (PAWP >15 mmHg, PVR >2 WU) Scleroderma has an annual prevalence of one to five cases for every 1000 individuals and nearly 15 percent of all cases develop PAH. A diagnosis of PAH in Scleroderma is virtually a death sentence, with studies reporting a mortality rate of 50 per cent in the 3 years of diagnosis. Therefore, developing and implementing screening and diagnosis protocol is important in the fight against this disease. echocardiography as the leading screening tool for scleroderma -PAH. In particular, systolic pulmonary arterial pressure (sPAP) and tricuspid regurgitation velocity (TRV). Echocardiography is non invasive tool for eary screening in pulmonary hypertension according ESC-ERS guideline If the peak tricuspid regurgitation velocity (TRV) is ≤ 2.8 m/s or not measurable, and there are no other echocardiographic signs of pulmonary hypertension, the probability is low.

If the TRV is ≤ 2.8 m/s or not measurable, but other echocardiographic signs of pulmonary hypertension are present, the probability is intermediate low

If the TRV is between 2.9 and 3.4 m/s and no other signs are present, the probability is intermediate high

If the TRV is between 2.9 and 3.4 m/s and other signs are present, the probability is high.

PH probability LOW → other causes . PH probability ntermediate low → follow up Echocardiography PH probability INTERMEDIATE high or HIGH → right heart catheterization Additional echocardiographic signs suggestive of pulmonary hypertension

A: The ventricles

RV/LV basal diameter area ratio ≥1.0

Flattening of the interventricular septum (LVEI >1.1 in systole and/or diastole)

TAPSE / sPAP ratio <0.55 mm/mmHg

B: Pulmonary artery

RVOT AT <105 ms and/or mid-systolic notching

Early diastolic pulmonary regurgitation velocity >2.2 m/s

PA diameter >25 mm

RPA diameter >25 mm

C: Inferior vena cava and RA

IVC diameter >21 mm with decreased inspiratory collapse (<50% with a sniff or <20% with quiet inspiration)

RA area (end-systole) >18 cm²

ELIGIBILITY:
Inclusion Criteria:

* . Inclusion criteria: aga ≥18 years confirmed diagnosis of scleroderma

Exclusion Criteria:

* aga <18 years
* patients refused to participate

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: aga ≥18 years confirmed diagnosis of scleroderma
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Screening for pulmonary hypertension in scleroderma patients | baseline
  detection rate of pulmonary hypertension in scleroderma by Echocardiography

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chennakesavulu PV, Uppaluri S, Koyi J, Jhaveri S, Avanthika C, Sakhamuri LT, Ashokbhai PK, Singh P. Pulmonary Hypertension in Scleroderma- Evaluation and Management. Dis Mon. 2023 Jul;69(7):101468. doi: 10.1016/j.disamonth.2022.101468. Epub 2022 Sep 24. PMID 36163292
- [Background] Kovacs G, Bartolome S, Denton CP, Gatzoulis MA, Gu S, Khanna D, Badesch D, Montani D. Definition, classification and diagnosis of pulmonary hypertension. Eur Respir J. 2024 Oct 31;64(4):2401324. doi: 10.1183/13993003.01324-2024. Print 2024 Oct. PMID 39209475
- [Background] Brown Z, Proudman S, Morrisroe K, Stevens W, Hansen D, Nikpour M. Screening for the early detection of pulmonary arterial hypertension in patients with systemic sclerosis: A systematic review and meta-analysis of long-term outcomes. Semin Arthritis Rheum. 2021 Jun;51(3):495-512. doi: 10.1016/j.semarthrit.2021.03.011. Epub 2021 Apr 4. PMID 33857705
- [Background] Chen K, See A, Shumack S. Epidemiology and pathogenesis of scleroderma. Australas J Dermatol. 2003 Feb;44(1):1-7; quiz 8-9. doi: 10.1046/j.1440-0960.2003.06301.x. PMID 12581091
- [Background] Humbert M, Kovacs G, Hoeper MM, Badagliacca R, Berger RMF, Brida M, Carlsen J, Coats AJS, Escribano-Subias P, Ferrari P, Ferreira DS, Ghofrani HA, Giannakoulas G, Kiely DG, Mayer E, Meszaros G, Nagavci B, Olsson KM, Pepke-Zaba J, Quint JK, Radegran G, Simonneau G, Sitbon O, Tonia T, Toshner M, Vachiery JL, Vonk Noordegraaf A, Delcroix M, Rosenkranz S; ESC/ERS Scientific Document Group. 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Heart J. 2022 Oct 11;43(38):3618-3731. doi: 10.1093/eurheartj/ehac237. No abstract available. PMID 36017548